CLINICAL TRIAL: NCT06056726
Title: Evaluation of Intra- and Peri-operative Complications and Disease-free Survival in Rectal Cancer Patients Undergoing Oncological Resective Surgery and Concomitant Bariatric Surgery
Brief Title: Evaluation of Surgical Complications and DFS in Obese Rectal Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Mario Musella MD, Full Professor of Surgery, Federico II University
Other Study IDs: RettOb
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Obesity, Morbid; Rectal Cancer; Surgery-Complications
Keywords: Bariatric Surgery; Oncological surgery
MeSH Terms: conditions — Obesity, Morbid; Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Obese Patients: Patients candidates for resective surgery for rectal cancer and also elegible for bariatric surgery
  Interventions: Procedure: BIB positioning

INTERVENTIONS:
Procedure: BIB positioning — BIB positioning in obese patients with rectal cancer elegible for neoadjuvant therapy

SUMMARY:
Obesity worsens treatment outcomes in rectal cancer patients: the local resective approach could in fact be more difficult in obese patients due to limited surgical visibility and it has also been reported that high visceral adiposity determines an increased risk of recurrence after chemoradiotherapy neoadjuvant. Bariatric surgery has proved to be the best choice for the treatment of morbid obesity and related comorbidities and in this context, the intragastric balloon (IGB) represents a strategy characterized by a low rate of complications and good results in terms of weight loss.

Therefore, the need to be able to offer obese patients suffering from rectal cancer the possibility of a better recovery perspective, alongside radical oncological surgery and neoadjuvant treatments, also a bariatric surgery such as the positioning of an intragastric balloon.

DETAILED DESCRIPTION:
Epidemiological data show that obesity is associated with a 30-70% increase in the risk of developing rectal cancer; Obesity could also be associated with a worsening of the tumor prognosis, with an increased risk of recurrence and increased mortality. From this point of view, recent studies have shown that a BMI ≥ 30 kg/m2 is associated with higher oncological and functional risks in patients with locally advanced rectal cancer, with lower response rates to neoadjuvant treatment and a less frequent preservation of the anal sphincter.

Obesity also worsens treatment outcomes: the local resective approach could in fact be more difficult in obese patients due to limited surgical visibility and it has also been reported that high visceral adiposity determines an increased risk of recurrence after chemoradiotherapy neoadjuvant. Bariatric surgery has proved to be the best choice for the treatment of morbid obesity and related comorbidities and in this context, the intragastric balloon (IGB) represents a strategy characterized by a low rate of complications and good results in terms of weight loss.

The most recent studies on the subject have shown that IGBs are effective in producing weight loss ranging from 6% to 15% compared to 1% -5% produced by lifestyle interventions alone Therefore, the need to be able to offer obese patients suffering from rectal cancer the possibility of a better recovery perspective (reduction of intra- and peri-operative complications, increased disease-free survival and lower risk of long-term recurrence) is underlined. ), alongside radical oncological surgery and neoadjuvant treatments, also a bariatric surgery such as the positioning of an intragastric balloon.

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally advanced rectal cancer in clinical stage II-III according to AJCC-UICC 2017 (candidates for neoadjuvant therapy)
* Patients suffering from I, II and III degree obesity at the same time
* Age between 18 and 70 years old
* BMI between 31 and 55 kg/m2
* Non-Smoking
* Candidates, according to AIOM guidelines, for rectal resection surgical procedures
* Candidates, according to SICOB guidelines, for an intragastric balloon placement procedure

Exclusion Criteria:

* Age ≤ 18 or ≥ 70 years
* BMI ≤ 30 or ≥ 59 Kg/m2
* Smoker
* Patients with non-locally advanced rectal cancer, not eligible for neoadjuvant therapy
* Histological positivity to Helicobacter pylori
* Presence of ulcerative lesions on EGD
* Previous bariatric surgery treatments

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese patients, with locally advanced rectal cancer in clinical stage II-III, candidates for neoadjuvant therapy, who can underwent BIB positioning during neoadjuvant period to obtain weight loss before resective cancer surgery
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2021-02-18 (Actual); Primary Completion 2024-02-18 (Estimated); Study Completion 2025-02-18 (Estimated)

PRIMARY OUTCOMES:
Peri-operative complications | Intra-operative complications and complications within 30 days from surgery
  Peri-operative complications during rectal cancer surgery

SECONDARY OUTCOMES:
Overall survival | 3 years after surgery
  Overall survival for patients with rectal cancer underwent resective surgery after BIB positioning

CONTACTS AND LOCATIONS:
Locations (1):
- Nunzio Velotti, Naples, Italy

IPD SHARING:
Plan to Share IPD: No